CLINICAL TRIAL: NCT07238348
Title: Prospective Evaluation of Analgesic Outcomes of Serratus Posterior Superior Intercostal Plane Block Versus Thoracic Epidural Analgesia and Systemic Opioid Analgesia After Video-Assisted Thoracoscopic Surgery
Brief Title: Analgesic Effectiveness of SPSIPB Versus Thoracic Epidural and Systemic Opioid Analgesia After VATS (SPSIPB-VATS)
Acronym: SPSIPB-VATS
Status: Not yet recruiting | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, Prof Dr, Karadeniz Technical University
Other Study IDs: 2024/176; 2024/276 (Other: Karadeiz Technical University, Local ethics Comitee)
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain Management; Video-assisted Thoracoscopic Surgery (VATS); Thoracic Epidural Analgesia; Serratus Posterior Superior Intercostal Plane Block
Keywords: Serratus Posterior Superior Intercostal Plane Block; Thoracic Epidural Analgesia; Systemic Opioid Analgesia; Video-Assisted Thoracoscopic Surgery; Opioid Consumption; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SPSIPB Group: Patients receiving Serratus Posterior Superior Intercostal Plane Block (SPSIPB) as part of routine postoperative analgesia for VATS.
- Thoracic Epidural Analgesia (TEA) Group: Patients receiving thoracic epidural analgesia with continuous epidural infusion for postoperative pain control following VATS.
- Systemic Opioid Analgesia Group: Patients managed with intravenous systemic opioid analgesia (e.g., tramadol PCA) as standard postoperative analgesia after VATS.

SUMMARY:
This prospective observational study aims to compare the postoperative analgesic effectiveness of three commonly used pain management strategies in video-assisted thoracoscopic surgery (VATS): Serratus Posterior Superior Intercostal Plane Block (SPSIPB), Thoracic Epidural Analgesia (TEA), and systemic opioid analgesia. The study evaluates postoperative pain scores, opioid consumption, and the need for rescue analgesics within the first 24 hours after surgery. By analyzing analgesic performance and safety profiles of these techniques, the study seeks to provide evidence to guide optimal postoperative pain management for patients undergoing minimally invasive thoracic procedures.

DETAILED DESCRIPTION:
This prospective observational clinical study investigates the comparative analgesic performance of three postoperative pain management strategies in patients undergoing video-assisted thoracoscopic surgery (VATS): Serratus Posterior Superior Intercostal Plane Block (SPSIPB), Thoracic Epidural Analgesia (TEA), and systemic opioid analgesia. SPSIPB is a recently defined interfascial plane block that may provide multi-dermatomal analgesia of the upper thoracic region with a less invasive profile compared with traditional neuraxial techniques. TEA, although considered effective for thoracic surgery, is associated with technical difficulty and potential adverse effects such as hypotension, urinary retention, and motor block. Systemic opioid analgesia remains widely used but may be limited by nausea, sedation, and opioid-related complications.

In this study, adult patients scheduled for elective VATS under general anesthesia will be managed with one of the three analgesic strategies as part of routine clinical practice. No randomization or allocation will be performed by the investigators; analgesic technique selection will follow standard clinical decision-making by the treating anesthesiologist. Postoperative pain will be evaluated using the Numerical Rating Scale (NRS) at predefined time points, including 0, 1, 2, 6, 12, and 24 hours after surgery. Total opioid consumption within the first 24 hours will be quantified as the primary outcome, expressed in tramadol-equivalent dosing. Secondary outcomes include the requirement for rescue analgesics, postoperative nausea and vomiting, hemodynamic parameters, and the Quality of Recovery-15 (QoR-15) score.

The study aims to provide comparative clinical evidence on the analgesic efficacy and tolerability of SPSIPB relative to TEA and systemic opioid analgesia in minimally invasive thoracic surgery. By identifying potential advantages or limitations of each technique, the findings may support optimization of multimodal analgesia protocols, improve postoperative comfort, and contribute to enhanced recovery strategies in VATS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years
* Scheduled for elective video-assisted thoracoscopic surgery (VATS)
* ASA physical status I-III
* Ability to understand study procedures and provide written informed consent
* Hemodynamically stable preoperatively

Exclusion Criteria:

* Known allergy or contraindication to local anesthetics or study medications
* Coagulopathy or use of anticoagulants not suitable for regional anesthesia
* Local infection or skin lesions at the injection site
* Severe pulmonary disease (e.g., severe COPD, uncontrolled asthma)
* Chronic opioid use or chronic pain disorders
* Neurological or psychiatric disorders impairing cooperation
* Pregnancy or breastfeeding
* BMI > 35 kg/m²
* Conversion from VATS to thoracotomy
* Inability to comply with postoperative assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-75 years) undergoing elective video-assisted thoracoscopic surgery (VATS) under general anesthesia at a tertiary university hospital. Patients will receive SPSIPB, thoracic epidural analgesia, or systemic opioid analgesia as part of routine clinical practice, and will be followed for postoperative pain outcomes within the first 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | 24 hours postoperatively
  Total Opioid Consumption at 24 Hours

SECONDARY OUTCOMES:
Pain Scores | 0, 1, 2, 6, 12, and 24 hours after surgery
  Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain.
Need for Rescue Analgesia | First 24 hours postoperatively
  Number of patients requiring additional analgesics despite standard postoperative analgesia.
Incidence of Postoperative Nausea and Vomiting (PONV) | First 24 hours postoperatively
  "PONV will be assessed using the Postoperative Nausea and Vomiting Intensity Scale (PONV Intensity Scale), which ranges from 0 to 3, where:
  0 = No nausea or vomiting
  1. = Mild nausea
  2. = Moderate nausea or single episode of vomiting
  3. = Severe nausea or two or more vomiting episodes
  Higher scores indicate more severe PONV. The presence of any nausea or vomiting and its severity will be recorded."
Heart Rate (beats per minute) | Intraoperative and first 24 hours postoperative
  "Heart rate will be recorded intraoperatively and during the first 24 postoperative hours. Heart rate is measured in beats per minute (bpm). Higher values indicate increased sympathetic activity or hemodynamic stress."
Quality of Recovery Score (QoR-15) | Preoperative baseline and 24 hours postoperative
  "The quality of postoperative recovery will be evaluated using the Quality of Recovery-15 (QoR-15) questionnaire.
  The QoR-15 is a validated patient-reported outcome measure with a score range from 0 to 150.
  0 = poorest possible recovery
  150 = best possible recovery
  Higher scores indicate better postoperative recovery. Scores will be recorded preoperatively (baseline) and at 24 hours postoperatively."
Time to First Opioid Request | First 24 hours postoperatively
  Time elapsed between arrival in the postoperative care unit and the first analgesic request via PCA.
Mean Arterial Pressure (mmHg) | Intraoperative and first 24 hours postoperative
  "Mean arterial pressure will be measured intraoperatively and during the first 24 postoperative hours. Mean arterial pressure is expressed in millimeters of mercury (mmHg). Higher or lower deviations from baseline may indicate hemodynamic instability."
Peripheral Oxygen Saturation (SpO₂,%) | Intraoperative and first 24 hours postoperative
  "Peripheral oxygen saturation (SpO₂) will be monitored intraoperatively and during the first 24 postoperative hours. SpO₂ is reported as a percentage (%), ranging from 0% to 100%, where higher values indicate better oxygenation."

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study does not include a data-sharing plan and contains identifiable clinical information that cannot be released.

REFERENCES:
- [Background] Bilal B, Ciftci B, Alver S, Ahiskalioglu A, Tulgar S. Serratus posterior superior intercostal plane block: novel block for minimal invasive cardiac surgery -A report of three cases. Korean J Anesthesiol. 2024 Feb;77(1):166-168. doi: 10.4097/kja.23542. Epub 2023 Oct 18. No abstract available. PMID 37852626
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Koksal BG, Baytar C, Bayraktar E, Balbaloglu H. Effects of serratus posterior superior intercostal plane block on postoperative analgesia in patients undergoing breast cancer surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Apr 24;25(1):209. doi: 10.1186/s12871-025-03092-0. PMID 40275145